CLINICAL TRIAL: NCT00258986
Title: Efficacy Study Comparing Hand-assisted Laparoscopic and Mini-incision Muscle Splitting Incision Living Donor Nephrectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UMCG/166.478/RvB
Record Dates: First submitted 2005-11-23; First posted 2005-11-28 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Living Donors
Keywords: Living donors; Nephrectomy; Kidney transplantation; Randomized Controlled Trial; Laparoscopy

INTERVENTIONS:
Procedure: Living donornephrectomy

SUMMARY:
The purpose of this study is to compare the effects of hand-assisted laparoscopic and mini-incision muscle-splitting donornephrectomy on living kidney donors. The hypothesis is that the mini-incision is not inferior to the laparoscopic technique.

DETAILED DESCRIPTION:
Living kidney donation has become an important source for kidney transplantation because of insufficient numbers of post mortem kidney donations. To reduce the surgical trauma of the donor operation and improve postoperative recovery minimal invasive techniques have developed. Especially the laparoscopic and the hand-assisted laparoscopic technique gained wide popularity. Minimal invasive open techniques have had less publicity. One of those open techniques is to perform the open donornephrectomy by means of an anterolateral approach. A transverse subcostal incision of 10 cm or less is made. The abdominal wall is opened by splitting the muscles and sparing the nerves. Staying in the retroperitoneal space the kidney is freed and taken out. Laparoscopic approaches have especially become more popular after the hand-assisted technique had developed. By means of an 8 cm transverse suprapubic skin incision and a vertical midline fascia incision the abdominal cavity is opened and a hand is inserted in the abdomen through an air tight sleeve. Three more trocarts are needed for the insufflation, the video camera and surgical instruments to perform a transperitoneal donornephrectomy. The hand in the abdomen assisting in the procedure has especially increased the sense of safety compared to the full laparoscopic technique without compromising the advantages of the laparoscopic technique.

So far no prospective or retrospective study has been done comparing the hand-assisted laparoscopic with the mini-incision muscle-splitting technique. Most studies that have been done comparing the (hand-assisted) laparoscopic technique with more invasive open techniques resulted in favour of the former technique.

Comparison(s): The study compares the effects of hand-assisted laparoscopic and mini-incision muscle-splitting donornephrectomy on living kidney donors.

ELIGIBILITY:
Inclusion Criteria:

* Accepted as living kidney donor by local protocol
* 18 years or older
* Excellent understanding of Dutch language
* Able to be operated on by both surgical techniques
* Having read patient information and signed informed consent

Exclusion Criteria:

* Previous surgery using subcostal incision(s)
* Not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Triple pain measurement using linear Visual Analogue Scale (at rest, at coughing and in supine position lifting of straight legs)

SECONDARY OUTCOMES:
- CRP levels in first three days after the donor operation (indicative of the magnitude of the surgical trauma)
- Abdominal wall muscle function (testing the functional integrity of the abdominal muscles)

CONTACTS AND LOCATIONS:
Overall Officials: Rutger J Ploeg, PhD, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Smit M, Hofker HS, Leuvenink HG, Krikke C, Jongman RM, Zijlstra JG, van Meurs M. A human model of intra-abdominal hypertension: even slightly elevated pressures lead to increased acute systemic inflammation and signs of acute kidney injury. Crit Care. 2013 Apr 4;17(2):425. doi: 10.1186/cc12568. No abstract available. PMID 23566574